CLINICAL TRIAL: NCT04850586
Title: The Impact of Structured Education Given by a Multidisciplinary Team on Pain, Anxiety, and Activities of Daily Living in Patients Undergoing Laparoscopic Cholecystectomy
Brief Title: Structured Education and Multidisciplinary Team
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Elif Gezginci, RN, PhD, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 45793301-604.01.01
Record Dates: First submitted 2021-04-18; First posted 2021-04-20 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Pain; Anxiety; Activities of Daily Living
Keywords: anxiety; cholecystectomy; education; multidisciplinary team; pain
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education Group (Experimental): The patients in the training group were given structured training by a multidisciplinary team. After the content of the structured education was prepared, three experts were consulted for their opinions in terms of the scope and content. Necessary adjustments were made in line with their recommendations. Patients in this group were visited in their rooms at least 12 hours before undergoing surgery by a multidisciplinary team consisting of a surgeon, an anesthesiologist, and a nurse. The multidisciplinary team visited the patients at the same time and provided their education after introducing the team. Structured verbal education and written documents were given to the patients for 30 minutes on preoperative preparation, anesthesia, intubation, mobilization, deep breathing and coughing exercises, nutrition and fluid management, the postoperative recovery process, clinical practice guideline and operating room protocols.
  Interventions: Other: Education Group
- Control Group (No Intervention): Routine education was given to the patients in the control group. Routine education was administered by a nurse working in the clinic after the patients were admitted to the hospital. The patients in this group were not trained by a multidisciplinary team. In the routine training, patients were only informed about preoperative preparation.

INTERVENTIONS:
Other: Education Group — The patients in the training group were given structured training by a multidisciplinary team. After the content of the structured education was prepared, three experts were consulted for their opinions in terms of the scope and content. Necessary adjustments were made in line with their recommendations. Patients in this group were visited in their rooms at least 12 hours before undergoing surgery by a multidisciplinary team consisting of a surgeon, an anesthesiologist, and a nurse. The multidisciplinary team visited the patients at the same time and provided their education after introducing the team. Structured verbal education and written documents were given to the patients for 30 minutes on preoperative preparation, anesthesia, intubation, mobilization, deep breathing and coughing exercises, nutrition and fluid management, the postoperative recovery process, clinical practice guideline and operating room protocols.
  Arms: Education Group

SUMMARY:
It is well-known that pre-operative education has a positive effect on patient recovery. This study was conducted to evaluate the impact of structured education given by a multidisciplinary team (surgeon, anesthesiologist, and nurse) on pain, anxiety, and activities of daily living in patients undergoing laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
In this randomized controlled study was conducted with 60 patients undergoing elective laparoscopic cholecystectomy in a training and research hospital in Turkey between March and August 2019. The participants were divided into two equal groups. Verbal structured education and written documents were given to the training group before surgery by a multidisciplinary team. The control group had the routine education. Data were collected using a Patient Information Form, the State Anxiety Inventory, a visual analog scale, and the Barthel Index for Activities of Daily Living.

ELIGIBILITY:
Inclusion Criteria:

* undergoing an elective laparoscopic cholecystectomy
* no loss of sensation related to vision and hearing
* opening to communication and cooperation
* no cancer diagnosis
* no chronic pain-related treatment
* no psychological disease diagnosis
* agreeing to participate in the study

Exclusion Criteria:

* undergoing emergency surgery
* hospitalized in the intensive care unit
* average score below 62 by Barthel Index

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-11-30 (Actual)

PRIMARY OUTCOMES:
The difference in pain scores measured by Visual Analog Scale between the two groups | The participants' pain levels were evaluated using the VAS at 06:00 AM on the first day of surgery.
  This scale is a unidimensional, valid and reliable scale in the measurement of acute pain intensity. This scale, which is comprised horizontally or vertically, consists of a 10 cm scale, at one end there is "no pain", at the other end there is "worst imaginable pain," with which the patient scores their pain. As the score on the scale increases, the severity of pain intensity increases.

SECONDARY OUTCOMES:
The difference in anxiety scores measured by State-Trait Anxiety Inventory between the two groups | Anxiety levels were evaluated using the STAI-I just before discharge (postoperative 1st day).
  The STAI measures two types of anxiety, state anxiety and trait anxiety. State Anxiety Inventory (STAI-I) is a sensitive tool for evaluating sudden changes in emotional reactions. It requires the individual to describe how they feel at a particular moment and under certain conditions and to respond by considering their feelings about the situation they are in. The scale consists of 20 items and the responses range from 1 to 4. The total score of the scale range from 20 to 80. High scores from the scale indicate high levels of anxiety and low scores indicate low levels of anxiety.
The difference in independence levels measured by the Barthel Daily Living Activities Index between the two groups | The independence levels of the patients in both groups were evaluated using the Barthel Daily Living Activities Index on the 10th-day follow-up appointment.
  This index consists of 10 items (feeding, bathing, grooming, dressing, bowels, bladder, toilet use, transfers (e.g. bed to chair and back), mobility on level surfaces (e.g. stairs), and questions the physical competence of the individual. Each item (unable, needs help, independent) is scored between 0-15 and 0-20 indicates total dependency; 21-61 indicates severe dependency, 62-90 indicates moderate dependency, 91-99 indicates slight dependency, and 100 indicates independence.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Gezginci, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- Saglık Bilimleri Universitesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zelenikova R, Homzova P, Homza M, Buzgova R. Validity and Reliability of the Czech Version of the Amsterdam Preoperative Anxiety and Information Scale (APAIS). J Perianesth Nurs. 2017 Oct;32(5):429-437. doi: 10.1016/j.jopan.2016.03.007. Epub 2016 Dec 28. PMID 28938978
- [Background] Zemla AJ, Nowicka-Sauer K, Jarmoszewicz K, Wera K, Batkiewicz S, Pietrzykowska M. Measures of preoperative anxiety. Anaesthesiol Intensive Ther. 2019;51(1):64-69. doi: 10.5603/AIT.2019.0013. PMID 31280554
- [Background] Lee CH, Liu JT, Lin SC, Hsu TY, Lin CY, Lin LY. Effects of Educational Intervention on State Anxiety and Pain in People Undergoing Spinal Surgery: A Randomized Controlled Trial. Pain Manag Nurs. 2018 Apr;19(2):163-171. doi: 10.1016/j.pmn.2017.08.004. Epub 2017 Nov 15. PMID 29153299
- [Background] Allvin R, Ehnfors M, Rawal N, Idvall E. Experiences of the postoperative recovery process: an interview study. Open Nurs J. 2008;2:1-7. doi: 10.2174/1874434600802010001. Epub 2008 Jan 4. PMID 19319214
- [Background] Pedziwiatr M, Mavrikis J, Witowski J, Adamos A, Major P, Nowakowski M, Budzynski A. Current status of enhanced recovery after surgery (ERAS) protocol in gastrointestinal surgery. Med Oncol. 2018 May 9;35(6):95. doi: 10.1007/s12032-018-1153-0. PMID 29744679
- [Background] Craig-Schapiro R, DiBrito SR, Overton HN, Taylor JP, Fransman RB, Haut ER, Sacks BC. Meet your surgical team: The impact of a resident-led quality improvement project on patient satisfaction. Am J Surg. 2018 Oct;216(4):793-799. doi: 10.1016/j.amjsurg.2018.07.056. Epub 2018 Aug 27. PMID 30177240
- [Background] Meissner W, Coluzzi F, Fletcher D, Huygen F, Morlion B, Neugebauer E, Montes A, Pergolizzi J. Improving the management of post-operative acute pain: priorities for change. Curr Med Res Opin. 2015 Nov;31(11):2131-43. doi: 10.1185/03007995.2015.1092122. Epub 2015 Sep 30. PMID 26359332
- [Background] Zieren J, Menenakos C, Mueller JM. Does an informative video before inguinal hernia surgical repair influence postoperative quality of life? Results of a prospective randomized study. Qual Life Res. 2007 Jun;16(5):725-9. doi: 10.1007/s11136-007-9171-y. Epub 2007 Feb 8. PMID 17286194
- [Background] Wongkietkachorn A, Wongkietkachorn N, Rhunsiri P. Preoperative Needs-Based Education to Reduce Anxiety, Increase Satisfaction, and Decrease Time Spent in Day Surgery: A Randomized Controlled Trial. World J Surg. 2018 Mar;42(3):666-674. doi: 10.1007/s00268-017-4207-0. PMID 28875242
- [Background] Diez-Alvarez E, Arrospide A, Mar J, Alvarez U, Belaustegi A, Lizaur B, Larranaga A, Arana JM. [Effectiveness of pre-operative education in reducing anxiety in surgical patients]. Enferm Clin. 2012 Jan-Feb;22(1):18-26. doi: 10.1016/j.enfcli.2011.09.005. Epub 2011 Dec 7. Spanish. PMID 22154548